CLINICAL TRIAL: NCT00994825
Title: Levosimendan to Reduce Mortality in High Risk Cardiac Surgery Patients. A Multicentre Randomized Controlled Trial
Brief Title: Levosimendan in High Risk Patients Undergoing Cardiac Surgery
Acronym: CHEETAH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, Head of Research, Anesthesia and Intensive Care Department, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GO/URC/ER/mm 768/DG
Record Dates: First submitted 2009-10-07; First posted 2009-10-14 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Low Cardiac Output Syndrome
Keywords: levosimendan; cardiac surgery; cardiac anesthesia; mortality; survival; inotropic drugs
MeSH Terms: conditions — Cardiac Output, Low | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): "Soluvit" ATC BO5XC (a mixture of vitamins with a yellow colour that is indistinguishable from the study drug Levosimendan) half ampul in 100 ml of glucose 5%
  Interventions: Drug: placebo
- Levosimendan (Experimental): Levosimendan
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan
  Other Names: simdax
  Arms: Levosimendan
Drug: placebo — "Soluvit" ATC BO5XC (a mixture of vitamins with a yellow colour that is indistinguishable from the study drug Levosimendan) half ampul in 100 ml of glucose 5%
  Arms: Placebo

SUMMARY:
Low cardiac output syndrome (LCOs) is a serious complication in critically ill patients or those undergoing major surgery, resulting in multiple organ damage with significant in-hospital and long-term morbidity and mortality, as well as prolonged hospital stay. In this setting the mortality rate is distressingly high despite improvements in intensive care treatment, but survivors have an acceptable quality of life.

DETAILED DESCRIPTION:
Low cardiac output syndrome (LCOs) is a serious complication in critically ill patients or those undergoing major surgery, resulting in multiple organ damage with significant in-hospital and long-term morbidity and mortality, as well as prolonged hospital stay. In this setting the mortality rate is distressingly high despite improvements in intensive care treatment, but survivors have an acceptable quality of life.

No inotropic drug has ever demonstrated to have beneficial effects on outcome in the setting of heart failure or in the perioperative period of major surgery. Previous studies and meta-analysis suggested an increased mortality in patients receiving "old" inotropic drugs. The originality of this large multicentre randomized placebo-controlled trial stands on the current non-evidenced-based-medicine use of inotropic agents in critically ill patients with low cardiac output syndrome or with decompensated heart failure.

Interestingly, the calcium sensitizer levosimendan has a double mechanism of action that could explain, in part, why do we expect to document, for the first time, a beneficial effect of an inotropic agent in clinically relevant outcomes: by binding to cardiac troponin C, it enhances myofilament responsiveness to calcium, thereby increasing myocardial contraction without increasing myocardial oxygen consumption; in addition, levosimendan activates adenosine triphosphate-dependent potassium channels which are important mediators of ischemic and pharmacological cardioprotection.

Most importantly, the originality of this trial will stay in the updated knowledge of the principal investigators. After publishing a first meta-analysis on this topic and documenting the cardioprotective properties of this drug, we performed further meta-analyses, and documented, for the first time, the possible beneficial effects on survival of an inotropic agent. Even if we presented the preliminary results of this meta-analysis to an important congress, we still have a "competitive advantage" with regard to other investigators who are not fully aware of the important results of these meta-analyses.

In the first meta-analysis a total of 139 patients undergoing cardiac surgery (5 randomized clinical trials) were randomized to receive levosimendan or best available treatment. We observed that levosimendan was associated with a significant reduction in cTn peak release (weighted mean difference = 2.5 ng/dl [-3.86,-1.14], p = 0.0003.) and in time to hospital discharge (weighted mean difference = -1.38 days [-2.78,0.03], p = 0.05).

The second, more updated meta-analysis (a total of 440 patients from 10 randomized controlled studies) was also performed in the specific setting of cardiac surgery. Levosimendan was associated with a significant reduction in postoperative mortality (11/235 [4.7%] in the levosimendan group vs 26/205 [12.7%] in the control arm, OR=0.38 [0.19-0.76], p for effect=0.007, NNT=12).

In the third meta-analysis, that included 3350 cardiac surgery and heart failure patients receiving levosimendan (1893 patients) or best available treatment (1457 patients) the use of levosimendan was associated with a significant reduction in mortality (333/1893 [17.6%] in the levosimendan group vs 326/1457 [22.4%] in the control arm, OR=0.74 [0.62-0.89], p for effect=0.001 NNT=21).

It should be underlined that no inotropic drug has ever demonstrated to have beneficial effects on outcome in the setting of heart failure or cardiac surgery. On the contrary, previous studies and meta-analysis suggested an increased mortality in patients receiving "old" inotropic drugs.

Study hypothesis is that levosimendan can reduce mortality in high risk patients undergoing cardiac surgery

It should be underlined that we're planning to treat patients "early" in the course of their low cardiac output syndrome: at the beginning of surgery in case of an ejection fraction< 25%, immediately after cardiopulmonary bypass in those patients who need high doses inotropic drugs for weaning, and early in the intensive care in those patients who will develop an initial low cardiac output syndrome within 24 hours from surgery).

In summary, the originality of this study includes:

* studying a clinical setting with an high mortality rate where all previously studied inotropic agents have failed
* using updated evidence based medicine (meta-analyses) as background and study hypothesis

  * involving those patients who would benefit more from cardiac protection (those with an early low cardiac output syndrome)
  * using a new inotropic agents that does not increase myocardial oxygen consumption and that have pharmacological preconditioning effects According to a recent meta-analysis, (1) the use of levosimendan reduces mortality in cardiac surgery. Common experience and further meta-analyses also suggest that the beneficial cardioprotective effects of this agent could also translate into a reduced intensive care and hospital stay. This will likely result in a decrease in the use of hospital resources and, therefore, in the cost of care. This effect will be important because we will selectively enroll high risk patients in which the risk of death is very high. Reduction in cost per patient will be also relevant.

The aim of this randomised, double blind study is to confirm the promising results of the above cited meta-analyses and to provide valid clinical evidence on the properties of levosimendan in critically ill patients undergoing cardiac surgery.

30.000 cardiac surgical interventions are performed in Italy every year (and 1.000.000 in the world). Since mortality in 2% of the general population and up to 20% in high risk subgroups, we estimate that up to 150 high risk patients per year and 100 low risk patients (overall 7.500 in the world) could benefit (survive) yearly thanks to the results of this study.

Reduction in cost per patient will be striking, since low cardiac output syndrome prolongs intensive care and hospital stay.

Study procedures We're planning a large randomized double-blind clinical trial (levosimendan vs placebo) that will enroll patients undergoing cardiac surgery (such as coronary artery bypass grafting, valvular repair or replacement, ascending aorta replacement…).

The study drug will be administered in the Intensive Care Unit for 24-48 hours and the patients observed till ICU discharge. Telephone follow up will be performed at 30 days and at one year.

Randomization Subjects will be allocated according to a centralized randomization derived from a computer-generated list of random number (in a sealed opaque envelope) that will be available only shortly before the preparation of the study drug. Data will be collected by trained observers who will not participate in patient care and will be blinded to the administered drug. The randomisation, performed at the last available moment, will reduce most biases together with the double blindness of the study.

The study will be conducted in cardiac surgery operating rooms and intensive care units of Italian Teaching Hospital. This hospitals have the structure and equipment to conduct the research. It should be underlined that the study has a very simple design and that the administration of levosimendan versus placebo will be the only non-routinely part of the management of the enrolled patients. All the patients included in the study will be strictly assisted by qualified personnel evaluating all the possible clinical variations. All of them will be routinely and invasively monitored.

According to the literature, Levosimendan will be administered at a starting dose of 0.05 ug/kg/min (ranging from 0.05 to 0.2 ug/kg/min) for 24-48 hours (or till discharge from the intensive care unit). Levosimendan will be diluted as follows: 1 ampul of 5 ml (2.5 mg/ml) in 100 ml of glucose 5%. Levosimendan will be compared in a double blind randomised fashion to placebo prepared as follows: "Soluvit" ATC BO5XC (a mixture of vitamins with a yellow colour that is indistinguishable from the study drug Levosimendan) half ampul in 100 ml of glucose 5% Both Levosimendan and placebo (soluvit) will be kept in fridge. The study drug will be started in the operating room or in ICU.

The drug is safe and has been administered to thousands of patients in the last few years. The patients included in this protocol are high risk patients undergoing cardiac surgery. We planned to notify to the Ministry any adverse reaction directly related to the drug and to the Hospital authorities all the observed death. The complications (adverse events) that commonly occur after cardiac surgery will be considered "disease progression" and will not be reported to the authorities during the study, but will be promptly available and will be listed in the results of the final manuscript.

The patients included in this study will receive a standard intensive treatment (general anesthesia, pacing, inotropic drugs, mechanical ventilation, postoperative sedation, diuretics, intravenous fluids, antibiotics….) monitoring (invasive arterial pressure, electrocardiogram, central venous pressure, pulseoximetry, temperature, arterial blood gases) and frequent routinely laboratory examination. All patients will receive a standard premedication, will have one large-bore iv catheter and a radial artery cannulated before induction of anaesthesia; pulse oximetry, 5 leads ECG with automated ST-segment analysis, central venous pressure, capnometry and urine output will be monitored as well. Temperature will be monitored with a bladder or rectal probe. Transesophageal echocardiography will be used at CPB weaning for clinical purposes, but the data will not be recorded. Induction of anaesthesia will be performed with ipnotic and analgesics and orotracheal intubation facilitated by muscle relaxants. Anaesthesia will be maintained with intravenous or volatile agents. No aprotinin will be used. CPB will be conducted with institutional custom packs. Myocardial protection will be ensured by cardioplegia solutions. After surgery, patients will be transferred to the intensive care unit (ICU)and weaned from the ventilator as soon as they were hemodynamically stable with no major bleeding, normothermic, and adequate levels of consciousness and pain control will be achieved. Weaning from the catecholamine infusion will be guided by standard hemodynamic criteria. Postoperative pain relief will be provided to all patients.

Decision to transfer the patient from the ICU to the ward will be based on these criteria: SpO2 >94% at an FiO2 <0.5 by facemask, adequate cardiac stability with no hemodynamically significant arrhythmias, chest tube drainage <50 ml/h, urine output >0.5 ml/kg/h, no intravenous inotropic or vasopressor agent in excess of dopamine 5 ug/kg/min, and no seizure activity. Criteria for hospital discharge will be hemodynamic and cardiac rhythm stability, presence of clean and dry incisions, afebrile, normal bowel movement, and independent ambulation and feeding.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Perioperative myocardial dysfunction

Exclusion Criteria:

* Previous unusual response to levosimendan or soluvit or any of their components
* Inclusion in other randomised controlled studies in the previous 30 days
* Levosimendan administration in the previous 30 days
* Parkinson's disease
* Emergency operation
* Kidney or liver transplant
* Liver cirrhosis (Child B or C)
* Decision to use ECMO (ECMO already started or planned)
* Do not resuscitate patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mortality | 30-days

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zangrillo, MD, Study Chair — Vita-Salute University of Milano
Locations (18):
- Santa Casa de Misericórdia de Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil
- Italy (13):
  - Policlinico S.Orsola-Malpighi, Bologna, Italy
  - Azienda Ospedaliera Universitaria San Martino, Genova, Italy
  - Azienda Ospedaliera Ospedali Riuniti Papardo - Piemonte, Messina, ME
  - Azienda Ospedaliera Regionale San Carlo, Potenza, Potenza
  - Ospedale Civile SS Annunziata, Sassari, Sassari
  - A.O.U. Citta della Salute e della Scienza, Torino, TO
  - A. O. Ordine Mauriziano di Torino, Torino, TO
  - Ospedale San Bortolo, Vicenza, VI
  - Azienda Ospedaliera Universitaria "Mater Domini", Catanzaro
  - Ospedale San Raffaele di Milano, Italy, Milan
  - Ospedale San Gerardo di Monza, Monza
  - Azienda Ospedaliera Specialistica dei Colli, Napoli
  - Azienda Ospedaliera Universitaria Pisana, Pisa
- Russia (4):
  - Astrakhan Federal Centre for Cardiac Surgery, Astrakhan, Russia
  - Scientific Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo, Russia
  - Moscow Regional Clinical & Research Institute, Moscow, Russia
  - Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Background] Landoni G, Mizzi A, Biondi-Zoccai G, Bruno G, Bignami E, Corno L, Zambon M, Gerli C, Zangrillo A. Reducing mortality in cardiac surgery with levosimendan: a meta-analysis of randomized controlled trials. J Cardiothorac Vasc Anesth. 2010 Feb;24(1):51-7. doi: 10.1053/j.jvca.2009.05.031. Epub 2009 Aug 22. PMID 19700350
- [Background] Landoni G, Zambon M, Zangrillo A. Reducing perioperative myocardial infarction with anesthetic drugs and techniques. Curr Drug Targets. 2009 Sep;10(9):858-62. doi: 10.2174/138945009789108837. Epub 2009 Sep 1. PMID 19538174
- [Background] Zangrillo A, Biondi-Zoccai G, Mizzi A, Bruno G, Bignami E, Gerli C, De Santis V, Tritapepe L, Landoni G. Levosimendan reduces cardiac troponin release after cardiac surgery: a meta-analysis of randomized controlled studies. J Cardiothorac Vasc Anesth. 2009 Aug;23(4):474-8. doi: 10.1053/j.jvca.2008.11.013. Epub 2009 Feb 12. PMID 19217315
- [Background] Landoni G, Rodseth RN, Santini F, Ponschab M, Ruggeri L, Szekely A, Pasero D, Augoustides JG, Del Sarto PA, Krzych LJ, Corcione A, Slullitel A, Cabrini L, Le Manach Y, Almeida RM, Bignami E, Biondi-Zoccai G, Bove T, Caramelli F, Cariello C, Carpanese A, Clarizia L, Comis M, Conte M, Covello RD, De Santis V, Feltracco P, Giordano G, Pittarello D, Gottin L, Guarracino F, Morelli A, Musu M, Pala G, Pasin L, Pezzoli I, Paternoster G, Remedi R, Roasio A, Zucchetti M, Petrini F, Finco G, Ranieri M, Zangrillo A. Randomized evidence for reduction of perioperative mortality. J Cardiothorac Vasc Anesth. 2012 Oct;26(5):764-72. doi: 10.1053/j.jvca.2012.04.018. Epub 2012 Jun 20. PMID 22726656
- [Background] Landoni G, Biondi-Zoccai G, Greco M, Greco T, Bignami E, Morelli A, Guarracino F, Zangrillo A. Effects of levosimendan on mortality and hospitalization. A meta-analysis of randomized controlled studies. Crit Care Med. 2012 Feb;40(2):634-46. doi: 10.1097/CCM.0b013e318232962a. PMID 21963578
- [Derived] Zangrillo A, Lomivorotov VV, Pisano A, Calabro MG, Belletti A, Brazzi L, Grigoryev EV, Guarracino F, Monaco F, Garofalo E, Crivellari M, Likhvantsev VV, Fominskiy EV, Paternoster G, Yavorovskiy A, Pasyuga VV, Oriani A, Lembo R, Bianchi A, Scandroglio AM, Abubakirov MN, Di Tomasso N, Landoni G; CHEETAH Study Group. Long-term outcome of perioperative low cardiac output syndrome in cardiac surgery: 1-year results of a multicenter randomized trial. J Crit Care. 2020 Aug;58:89-95. doi: 10.1016/j.jcrc.2020.04.005. Epub 2020 Apr 17. PMID 32402931
- [Derived] Landoni G, Lomivorotov VV, Alvaro G, Lobreglio R, Pisano A, Guarracino F, Calabro MG, Grigoryev EV, Likhvantsev VV, Salgado-Filho MF, Bianchi A, Pasyuga VV, Baiocchi M, Pappalardo F, Monaco F, Boboshko VA, Abubakirov MN, Amantea B, Lembo R, Brazzi L, Verniero L, Bertini P, Scandroglio AM, Bove T, Belletti A, Michienzi MG, Shukevich DL, Zabelina TS, Bellomo R, Zangrillo A; CHEETAH Study Group. Levosimendan for Hemodynamic Support after Cardiac Surgery. N Engl J Med. 2017 May 25;376(21):2021-2031. doi: 10.1056/NEJMoa1616325. Epub 2017 Mar 21. PMID 28320259
- See also: italian association of cardiothoracic anesthesiologists — http://www.itacta.org
- See also: italian society of anesthesiologists — http://www.siaarti.it